CLINICAL TRIAL: NCT06303245
Title: Combined Effects of Abdominal Binders and TENS on Post-operative Pain, Distress and Constipation in Puerperium Period After Cesarean Section
Brief Title: Effects of Abdominal Binders and TENS on Puerperium Period After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0579
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Cesarean Section; Complications, Wound, Dehiscence
Keywords: Cesarean section; constipation; Post-operative pain; puerperium; TENS
MeSH Terms: conditions — Wounds and Injuries; Constipation; Pain, Postoperative | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABDOMINAL BINDERS (Experimental)
  Interventions: Other: ABDOMINAL BINDERS
- TENS (Active Comparator)
  Interventions: Other: TENS

INTERVENTIONS:
Other: ABDOMINAL BINDERS — will be given abdominal binders along with basic physiotherapy care. Physiotherapy care will include sitting exercises such as deep breathing exercises, protected huffing technique will be performed to improve gases exchange and remove secretion. In supine exercises such as basic ROM, ankle pumps, pelvic rolling, leg sliding will be performed. Each exercise will be of 10 repetition. This exercise will be given for 2 days per week for 6 weeks. Along with these exercises education related postural management and breastfeeding positions will also be guided
  Arms: ABDOMINAL BINDERS
Other: TENS — will receive TENS with high frequency (F=100Hz and T=100μs), intensity according to patient's pain threshold, duration of 30 continuous minutes, 2 cm above and below incision, with electrodes transversally positioned and crossing the incision. Two treatment sessions will be done per week for the period of 6 weeks. This group will be given tens along with abdominal binders with basic physiotherapy care. (23) In this treatment female's abdomen will be measured by a standard inch tape, then, according to the abdominal circumference, the binder will be fastened for 6 weeks. The binder will be placed tightly at the lower abdominal level with the incision positioned at the middle part of the binder. Participants will be asked to note the time to record the duration of binder wearing before taking the break. The binder will be opened between 10 pm and 8 am. This group will be given abdominal binders along with basic physiotherapy care
  Arms: TENS

SUMMARY:
To determine the combined effects of abdominal binders and TENS on post-operative pain, distress and constipation in puerperium period after cesarean section

ELIGIBILITY:
Inclusion Criteria:

* Participants on early puerperium period having constipation and willing to participate.
* Primigravida
* Body mass index (BMI) less than 30 kg/m2

Exclusion Criteria:

* Laxatives-induced patients
* History of chronic constipation
* Post cesarean abdominal suture infection.
* People with chronic diseases, and who underwent non-routine or additional surgical procedures, such as hysterectomy, tubal ligation, and classical uterine incision.
* Participants with inability to tolerate the binder.
* Participants who show unwillingness to participate in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — PUERPERIUM PERIOD AFTER CESAREAN SECTION
Enrollment: 50 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
o Numeric Pain rating Scale | 6th week
  Numeric pain rating scale is a subjective measure 11 point numerical scale which is used to measure pain. Is scoring range In this scale 0 shows no pain and 10 shows worst pain imaginable. It has good reliability of 0.79 and validity of 0.96.
o Symptom Distress scale | 6th week
  Symptom distress scale is a 13 item self-assessment scale with 13 symptoms like pain, fatigue, insomnia, lack of appetite, nausea, breathlessness, lack of concentration, lack of appetite and altered mood. It's scoring is done by using 5 point Likert scale where 1 shows least distress and 5 shows extreme distress. With a total score ranging from 13 to 65. It has a reliability of 0.821 and validity of 0.825.
o PAC-SYM Questionnaire | 6th week
  The PAC-SYM is a tool which is used to assess the severity of constipation. It range is from 0 and 48. Less value shows less severity of constipation. The patients were then asked to rate the severity of each symptom in a 5-point Likert scale (0-4; absent to very severe) during the past 2 weeks. The items were further categorized into 3 domains: abdominal symptoms (question 1-4), rectal symptoms (question 5-7), and stool symptoms (question 8-12). It is a reliable tool with value of 0.66 and validity with value of 0.75

CONTACTS AND LOCATIONS:
Overall Officials: hina gul gul, Principal Investigator — Riphah International University
Locations (1):
- PAF hospital and sheikh zayed hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira VB, Iuamoto LR, Hsing WT. Multidisciplinary management of musculoskeletal pain during pregnancy: A review of literature. Journal of the International Society of Physical and Rehabilitation Medicine. 2021;4(2):63-9.
- [Background] Wakkar A, Patil SP. Assessment of knee and ankle proprioception during the third trimester of pregnancy and postpartum period among primiparous women: An observational longitudinal study. J Educ Health Promot. 2022 Jul 29;11:241. doi: 10.4103/jehp.jehp_311_22. eCollection 2022. PMID 36177431
- [Background] Jenabi E, Khazaei S, Bashirian S, Aghababaei S, Matinnia N. Reasons for elective cesarean section on maternal request: a systematic review. J Matern Fetal Neonatal Med. 2020 Nov;33(22):3867-3872. doi: 10.1080/14767058.2019.1587407. Epub 2019 Mar 8. PMID 30810436
- [Background] Mohamed H, Yousef A, Kamel H-E, Oweda K, Abdelsameaa G. Kinesio taping and strength recovery of postnatal abdominal muscles after cesarean section. Egyptian Journal of Physical Therapy. 2020;4(1):13-9
- [Background] Verma V, Vishwakarma RK, Nath DC, Khan HTA, Prakash R, Abid O. Prevalence and determinants of caesarean section in South and South-East Asian women. PLoS One. 2020 Mar 12;15(3):e0229906. doi: 10.1371/journal.pone.0229906. eCollection 2020. PMID 32163440
- [Background] Kuronen M. Constipation and pain management after spine surgery and in pregnancy and postpartum: Itä-Suomen yliopisto; 2021.
- [Background] Orlova D. MODERN POSSIBILITIES FOR CORRECTING CONSTIPATION IN POSTPARTUM WOMEN. Молодежный инновационный вестник. 2021;10(S1):29-32.